CLINICAL TRIAL: NCT01183208
Title: A Phase I, Single-Centre, Double-Blind, Randomised, Placebo-Controlled, Parallel Group, Pharmacokinetic and Safety Study to Evaluate Systemic Exposure and Local Vaginal Exposure to Lidocaine and Prilocaine and the Metabolites 2,6 DiMethylAlanine (2, 6, DMA) and O-Toluidine; and the Safety and Tolerability of PSD502 in Female Healthy Volunteer Subjects Following Daily Application to the Vagina and Cervix for Seven Days With Three Different Doses of PSD502 or Placebo
Brief Title: A Safety and Tolerability Study of Administration of PSD502
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Plethora Solutions Ltd (Industry)
Collaborators: Bio-Kinetic Europe, Ltd. (Industry); Omnicare Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSD502-PE-006
Record Dates: First submitted 2010-01-26; First posted 2010-08-17 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 active treatment and placebo (Experimental): Active treatment and placebo
  Interventions: Drug: Intervention A; Drug: Intervention D
- Cohort 2 - Active treatment and placebo (Experimental): Active treatment and placebo
  Interventions: Drug: Intervention B; Drug: Intervention D
- Cohort 3 Active Treatment and placebo (Experimental): Active treatment and placebo
  Interventions: Drug: Intervention C; Drug: Intervention E

INTERVENTIONS:
Drug: Intervention A — A single dose of 3 mg will consist of 3 sprays of the 1 mg strength spray applied topically to cervix (1 spray) and vaginal fornices (2 sprays)
  Arms: Cohort 1 active treatment and placebo
Drug: Intervention B — A single dose of 30 mg will consist of 3 sprays of the 10 mg strength spray applied topically to cervix (1 spray) and vaginal fornices (2 sprays)
  Arms: Cohort 2 - Active treatment and placebo
Drug: Intervention C — A single dose of 150 mg will consist of 15 sprays of the 10 mg strength spray applied topically to cervix (5 sprays) and vaginal fornices (10 sprays)
  Arms: Cohort 3 Active Treatment and placebo
Drug: Intervention D — A dose of placebo will consist of 3 sprays of the placebo spray applied topically to cervix (1 spray) and vaginal fornices (2 sprays)
  Arms: Cohort 1 active treatment and placebo; Cohort 2 - Active treatment and placebo
Drug: Intervention E — A dose of placebo will consist of 15 sprays of the placebo spray applied topically to cervix (5 sprays) and vaginal fornices (10 sprays)
  Arms: Cohort 3 Active Treatment and placebo

SUMMARY:
A Phase I, Single-Centre, Double-Blind, Randomised, Placebo-Controlled, Parallel Group, Pharmacokinetic and Safety Study to Evaluate Systemic Exposure and Local Vaginal Exposure to Lidocaine and Prilocaine and the Metabolites 2,6 DiMethylAlanine (2, 6, DMA) and O-Toluidine; and the Safety and Tolerability of PSD502 in Female Healthy Volunteer Subjects Following Daily Application to the Vagina and Cervix for Seven Days With Three Different Doses of PSD502 or Placebo

DETAILED DESCRIPTION:
The study drug is a metered-dose anaesthetic spray, which is being developed for the treatment of premature ejaculation (PE). The use of anaesthetic in topical creams has been well established, and there is a licensed topical anaesthetic cream in the market with the same active ingredients as the spray (eutectic mixture of local anaesthetics cream 5%, lidocaine & prilocaine). The use of a cream does not result in the concentrated drug being in direct contact with the cells, unlike the spray.

Six clinical studies have already been carried out for the spray; two involved the recruitment of 556 PE patients with some being dosed for up to 1 year. These studies have demonstrated a prolongation of intravaginal ejaculatory latency time and no safety concerns for male patients or their female partners. The partners of clinical study participants have been asked to report health changes during the studies. Reports of vaginal numbness were uncommon; however, effects of the transfer to a partner cannot be excluded. This study is being conducted to determine the effects of the drug on the whole body in females as well as local vaginal exposure to the spray. This study will be conducted in order to support a marketing application in the United States (US) at the request of the U.S. Food and Drug Administration.

ELIGIBILITY:
Inclusion Criteria:

* Female non-smokers aged 18 years old and over
* Willing and able to provide written informed consent
* Generally, in good health in the opinion of the investigator
* Subject must have a body mass index between 18 and 30 kg/m2, inclusive
* Willing and able to comply with all study procedures in the opinion of the investigator
* Negative Papanicolaou smear performed either during gynaecological examination at screening or documented in the 12 months prior to study entry
* Negative drugs of abuse and cotinine test at screening
* Female subjects of child-bearing potential who are sexually active or become sexually active must be using a method of effective contraception from 14 days before screening and continue to use this until the end of the study (If oral contraceptives are used, these must have been stable for a period of 3 months. If a barrier method is being used, this should be latex based and not polyurethane based)
* Female subjects who are post-menopausal must have been post-menopausal >1 year and have confirmed elevated serum follicle stimulating hormone at screening

Exclusion Criteria:

* History of a significant medical condition that would preclude further study participation, in the opinion of the investigator
* Currently taking, or has taken within the 2 weeks prior to screening, any concomitant medication that could confound interpretation of the safety or pharmacokinetic data on PSD502. Use of prescription medication within 14 days or over-the-counter products within 7 days prior to first dose
* Suffering from an sexually transmitted disease, or is positive for hepatitis B, hepatitis C, or human immunodeficiency virus infection
* Safety testing: abnormalities at screening, in particular liver function tests, which are indicative of a medical condition and that would preclude further participation, in the opinion of the investigator
* Significant abnormality of the vaginal mucosa or cervix that would preclude interpretation of the examination of these areas or that could be worsened by use of PSD502
* History of alcohol or drug abuse within 1 year prior to screening
* Known drug sensitivity to amide-type local anaesthetics
* Unlikely to understand or be able to comply with study procedures, for any reason, in the opinion of the investigator
* History of glucose-6-phosphate dehydrogenase deficiency or use of medications that would increase susceptibility to methemoglobinemia (e.g., anti-malarial agents)
* Use of class I (e.g., mexiletine, tocainide) and III (e.g., amiodarone, sotalol) anti-arrhythmic drugs
* Subject has received an investigational (non-registered) drug within 90 days of screening
* Subject has any physical or psychological condition that would prevent them from undertaking the study procedures, including, but not limited to, the following:

  * Uro-gynaecological disease or recent surgery within 8 weeks of screening which would make intravaginal application or vaginal examination/colposcopy difficult or painful OR
  * Ongoing significant psychiatric disorder (e.g., bipolar disease, depression/anxiety disorder or schizophrenia)
* Subject has a clinically obvious vaginal infection, such as active vaginal Candida albicans (thrush), or other abnormal vaginal discharge
* Subjects who are pregnant or lactating
* Subjects should not be menstruating during the treatment phase
* Subjects who refuse to allow their primary care physician to be informed of their participation
* Donation of blood or blood products within 90 days prior to dosing or at any time during the study, except as required by this protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of adverse events, serious adverse events, findings from the examination of the cervix and vagina, vital signs, electrocardiogram data, hematology, and biochemistry parameters | Throughout the study

SECONDARY OUTCOMES:
Pharmacokinetic parameters: AUC0-t, AUC0-inf, AUCtau, Rc, Cmax, tmax, t½ and kel | Days 1 through 7
Vaginal fluid analysis for active ingredients and metabolites | Days 2 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (1):
- Bio-Kinetic Europe Limited, Belfast, United Kingdom